CLINICAL TRIAL: NCT00200733
Title: The Use of Narrative in Public Health Research and Practice: Patient Experience of Wellness Acupuncture
Status: Terminated | Type: Observational
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Other Study IDs: F31AT000789-01 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2005-12

CONDITIONS: Pain; Depression; Fatigue
Keywords: acupuncture; patient narratives; qualitative methods
MeSH Terms: conditions — Pain; Depression; Fatigue

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study examined the experiences of individuals undergoing acupuncture to gather information on patient-provider communication and on the therapeutic effects of acupuncture.

DETAILED DESCRIPTION:
Authentic voice is a approach involving the use of first-hand narratives from members of a target population in order to accomplish public health goals. In the first paper, a discussion of the potential of using narratives from the target population as 1) a direct intervention; 2) a form of persuasive communications; and 3) a source of information for research into various topics. The main premise is that traditional narrative methods can be adapted to the public health context by providing the narrator with the topic of the narrative. The second paper examines the patient experience of acupuncture using narrative drawn from interviews with and letters from acupuncture patients using a content oriented approach. The third paper examines the importance of meaning shift over the course of acupuncture treatment and demonstrates the usefulness of patient narratives as a data source for examining meaning. Findings include the need for intervention studies comparing authentic voice approaches to existing health communication tools for effectiveness in creating attitude and behavior change efficiently. Authentic voice approaches also need to be researched to understand and systematize concepts such as validity in relation to target-group derived narratives. Effectiveness of authentic voice for advocacy and research should also be further tested. Concerning acupuncture, the second and third papers show that acupuncture patients report a variety of benefits far wider than previously reported in the literature. Study designs should consider this wide range of benefits when assessing acupuncture outcome. Meaning shift is also reported by acupuncture patients and may play an important (but non-specific) role in the healing associated with acupuncture.

ELIGIBILITY:
Inclusion Criteria:

* individuals seeking acupuncture from private practice in Baltimore/Washington metro area.

Exclusion Criteria:

* prior patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2003-06; Study Completion 2004-03

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Stibich, PhD, Principal Investigator — Johns Hokins School of Public Health